CLINICAL TRIAL: NCT06640673
Title: Electrophysiological Signature of Mild Cognitive Impairment and Its Relationship with Parkinson's Disease: a High-density EEG Investigation
Acronym: MMCI
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 2023.06
Record Dates: First submitted 2024-02-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease; Parkinson Disease, Mild Cognitive Impairment; Healthy
Keywords: MCI in PD; Mild Cognitive Impairment; Parkinson's disease; Hd-EEG
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PD-MCI: Parkinson's disease with Mild Cognitive Impairment
  Interventions: Diagnostic Test: Hd-EEG
- PD-nMCI: Parkinson's disease without Mild Cognitive Impairment
  Interventions: Diagnostic Test: Hd-EEG
- Healthy control: Healthy participants matched for age and gender with the experimental groups
  Interventions: Diagnostic Test: Hd-EEG

INTERVENTIONS:
Diagnostic Test: Hd-EEG — Subjects undergo a clinical and neuropsychological assesment, then a Hd-EEG both during resting state and execution of tasks, and structural Magnetic Resonance Imaging
  Other Names: MRI

SUMMARY:
The study aims to investigate neural correlate of Mild Cognitive Impairment (MCI) in Parkinson's disease (PD) and to identify a link between functional impairment (in both cognitive and motor domains) and electrophysiological cortical sing of MCI in PD. A sample of 42 subjects will be divide into three subgroup: healthy control, PD with MCI (PD-MCI) and PD without MCI (PD-ctrl). Those subjects will undergo a specific neuropsychological evaluation and, to measure the electro-cortical activity, high-density electroencephalography (hdEEG) will be record during both resting state and cognitive tasks. Furthermore, hdEEG data will be combine with structural magnetic resonance to obtain information about network connectivity.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder, characterized by a degeneration of dopaminergic neurons at the level of the pars compacta of the substantia nigra, which results in impaired control of the nigrostriatal pathway. This degeneration is manifested by both motor and non-motor symptoms such bradykinesia, tremor, rigidity, and cognitive disorders. Particularly, patients with PD might be affected by Mild Cognitive Impairment (MCI), dementia, and related behavioral disorders including apathy and depressive syndromes. However, while motor disturbances are more evident, it is difficult to evaluate the onset of cognitive symptoms, especially in the prodromal phases of the disease. Indeed, it seems that the onset of cognitive deficits in PD occurs in a high prevalence in the earlier stages of the disease. PD patients can often be associated with MCI, a preclinical condition characterized by the presence of deficits in memory and executive functions as well as, to a lesser extent, in language- and visuospatial- related functions.

Dual-syndrome hypothesis posit the existence of two subtypes of MCI one fronto-striatal, characterised by executive and attentional deficits, and a posterior cortical one, characterised by deficits in memory visuo-spatial and language deficits. Recent studies described alterations in brain rhythm, measured with high-density EEG (HDEEG) in terms of frequency domain analysis, at the level of fronto-striatal regions only in patients with the fronto-striatal subtype. Moreover, fMRI studies have shown that the presence of MCI in PD causes a reduction in activity at the level of the cognitive cortico-striatal loop, which includes the caudate nucleus (CN) and prefrontal cortex (PFC).

Although the use of neurophysiological and neuroimaging techniques have substantially grown, the available data highlight the lack of detailed descriptions of functional connectivity in relation whit the onset and extent of the cognitive deficit itself. Therefore, the aim of the present study is to characterise MCI in PD from a neurophysiological and clinical point of view. First, all patients undergo a neuropsychological assessment to identify PD patients with MCI (PD-MCI) and those without MCI (PD-nMCI). Then, to investigate the functional connectivity of cortical areas underpinning cognitive decline, HDEEG will be record, during both resting state and cognitive tasks. Furthermore, for each participant will be collect MRI (Magnetic resonance imaging), to combine structural data with electrodes position over the scalp. This would allow obtaining a realistic model of the head for source analysis.

Identification of alterations in functional connectivity between specific cortical areas in MCI-PD patients, and a possible direct relationship between these and clinical impairment, could lead to improve therapeutic interventions and prevent cognitive disorders in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Upper score >24 MMSE or >15.5 Moca
* If taking medications, taking stable doses for at least 4 weeks prior to the inclusion visit - of anticholinesterase drugs (donepezil, memantine, rivastigmine, ...) or antidepressants (SSRIs, tricyclics, SNARI, ...) or Levodopa.
* Having signed the informed consent

Exclusion Criteria:

* Subjects with severe dementia ( MMSE < 24 )
* Lower score <15.5 Moca
* Subjects on antipsychotic treatment for less than 3 months
* Subjects with uncontrolled comorbidities
* Subjects with metal prostheses or dentures and in general conditions for which MRI examinations are prevented.
* Subjects with an inability to walk independently.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients will be recruited in the IRCCS San Camillo Hospital or through collaborators of the responsible researchers.
  Healty controls will be enrolled voluntarily.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2023-06-18 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Power Spectrum Density Analysis profile for hdEEG resting state data | at baseline
  For all the groups, starting from the hdEEG data, brain oscillation will be studied by performing the Power Spectral Analysis (PSD). The PSD aims to investigate the spectral properties in the delta (1-4 Hz), theta (4-8 Hz), alpha (8-13 Hz), beta (13-30 Hz), and gamma (>30Hz) frequencies bands. PSD will be performed for each electrode, for each subject, and then averaged across subjects, obtaining a value of PSD for each electrode, separately for each group (PD-ctrl vs PD-MCI). Then the PSD value will be displayed over the scalp with a topological representation.
Power Spectrum Density Analysis profile for hdEEG during cognitive task data | at baseline
  For all the groups, starting from the hdEEG data, brain oscillation will be studied by performing the Power Spectral Analysis (PSD). The PSD aims to investigate the spectral properties in the delta (1-4 Hz), theta (4-8 Hz), alpha (8-13 Hz), beta (13-30 Hz), and gamma (>30 Hz) frequencies bands. PSD will be performed for each electrode, for each subject, and then averaged across subject obtaining value of PSD for each electrode, separately for each group (PD-ctrl vs PD-MCI). Then the PSD value will be displayed over the scalp with a topological representation.
Functional connectivity - seed based analysis for hdEEG resting state data | at baseline
  To study the temporal correlation of cortical signals generated in spatially distributed regions of interest (ROI), the collected hdEEG data will be analyzed using the seed-based functional connectivity analysis (FC-SBA). FC-SBA will measures the time course activation of specific resting state networks (RSNs). Specifically, the DMN (default mode network), SN (Salience Network), FPN1 and FNP2 (Fronto-parietal Network). This approach allows to obtain the functional connectivity matrices that will show the activation pattern of different RSNs and frequency bands (delta 1-4Hz; theta 4-8Hz; alpha 8-13 Hz, beta 13-30Hz; gamma >30Hz).
Functional connectivity - seed based analysis for hdEEG during cognitive task data | at baseline
  To study the temporal correlation of cortical signals generated in spatially distributed regions of interest (ROI), the collected hdEEG data will be analyzed using the seed-based functional connectivity analysis (FC-SBA). FC-SBA will measures the time course activation of specific resting state networks (RSNs). Specifically, the DMN (default mode network), SN (Salience Network), FPN1 and FNP2 (Fronto-parietal Network). This approach allows to obtain the functional connectivity matrices that will show the activation pattern of different RSNs and frequency bands (delta 1-4Hz; theta 4-8Hz; alpha 8-13 Hz, beta 13-30Hz; gamma >30Hz).

SECONDARY OUTCOMES:
Performances at neuropsychological evaluation | at baseline
  Cognitive performances will be assessed before hdEEG by a neuropsychological battery encompassing the main cognitive domains. Specific neuropsychological tests will be administered according to the specific guideline for the cognitive evaluation in Parkinson's Disease, defined by the MDS Task Force.
  Raw scores at each test will be converted in z-scores based on each test normative data. Z-scores will be averaged to calculate composite scores for each cognitive domain. The composite scores will be the following: general cognitive functioning, attention, executive function, short-term memory, long-term memory, visuospatial abilities, language.
Fraility assessment | at baseline
  FRIED PHENOTYPE (PASE) analyzes 5 dimensions: presence of fatigue, grip strength, walking speed, unintentional weight loss, and level of activity. If at least 3 of these dimensions are deficient, then the patient is classified as frail; if 2 are deficient, the patient is pre-frail; if none are deficient, the patient is robust.
Accuracy during cognitive task | at baseline
  Accuracy during cognitive task will be extracted from the behavioral responses of each participant as the percentage of the correct responses. The accuracy at the task will be used as an additional parameter for analysis of the primary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: francesca burgio, phd, Principal Investigator — San Camillo IRCCS
Locations (1):
- IRCCS San Camillo S.R.L, Lido, Italy, Italy

REFERENCES:
- [Background] Nagano-Saito A, Habak C, Mejia-Constain B, Degroot C, Monetta L, Jubault T, Bedetti C, Lafontaine AL, Chouinard S, Soland V, Ptito A, Strafella AP, Monchi O. Effect of mild cognitive impairment on the patterns of neural activity in early Parkinson's disease. Neurobiol Aging. 2014 Jan;35(1):223-31. doi: 10.1016/j.neurobiolaging.2013.06.025. Epub 2013 Aug 7. PMID 23932879
- [Background] Betrouni N, Devignes Q, Bayot M, Derambure P, Defebvre L, Leentjens AF, Delval A, Dujardin K. The frontostriatal subtype of mild cognitive impairment in Parkinson's disease, but not the posterior cortical one, is associated with specific EEG alterations. Cortex. 2022 Aug;153:166-177. doi: 10.1016/j.cortex.2022.04.015. Epub 2022 May 11. PMID 35667287
- [Background] Monchi O, Petrides M, Doyon J, Postuma RB, Worsley K, Dagher A. Neural bases of set-shifting deficits in Parkinson's disease. J Neurosci. 2004 Jan 21;24(3):702-10. doi: 10.1523/JNEUROSCI.4860-03.2004. PMID 14736856
- [Background] Samogin J, Marino M, Porcaro C, Wenderoth N, Dupont P, Swinnen SP, Mantini D. Frequency-dependent functional connectivity in resting state networks. Hum Brain Mapp. 2020 Dec 15;41(18):5187-5198. doi: 10.1002/hbm.25184. Epub 2020 Aug 25. PMID 32840936
- [Background] Cai M, Dang G, Su X, Zhu L, Shi X, Che S, Lan X, Luo X, Guo Y. Identifying Mild Cognitive Impairment in Parkinson's Disease With Electroencephalogram Functional Connectivity. Front Aging Neurosci. 2021 Jul 1;13:701499. doi: 10.3389/fnagi.2021.701499. eCollection 2021. PMID 34276350
- [Background] Cera N, Esposito R, Cieri F, Tartaro A. Altered Cingulate Cortex Functional Connectivity in Normal Aging and Mild Cognitive Impairment. Front Neurosci. 2019 Sep 13;13:857. doi: 10.3389/fnins.2019.00857. eCollection 2019. PMID 31572106
- [Background] Gorges M, Muller HP, Lule D; LANDSCAPE Consortium; Pinkhardt EH, Ludolph AC, Kassubek J. To rise and to fall: functional connectivity in cognitively normal and cognitively impaired patients with Parkinson's disease. Neurobiol Aging. 2015 Apr;36(4):1727-1735. doi: 10.1016/j.neurobiolaging.2014.12.026. Epub 2014 Dec 31. PMID 25623332
- [Background] Litvan I, Goldman JG, Troster AI, Schmand BA, Weintraub D, Petersen RC, Mollenhauer B, Adler CH, Marder K, Williams-Gray CH, Aarsland D, Kulisevsky J, Rodriguez-Oroz MC, Burn DJ, Barker RA, Emre M. Diagnostic criteria for mild cognitive impairment in Parkinson's disease: Movement Disorder Society Task Force guidelines. Mov Disord. 2012 Mar;27(3):349-56. doi: 10.1002/mds.24893. Epub 2012 Jan 24. PMID 22275317